CLINICAL TRIAL: NCT00754806
Title: Prospective Randomized Study Between Open and Hand Assisted Splenectomies
Brief Title: Prospective Randomized Comparison of Clinical Results of Hand Assisted Laparoscopic Splenectomies and Open Splenectomies
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Istanbul Faculty of Medicine, Department of General Surgery
Other Study IDs: 1687-2007
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Postoperative Pain
Keywords: HALS; open splenectomy; splenomegaly; HALS as a hybrid approach of pure laparoscopy and open surgery has some definite advantages over open surgery; In the HALS group, incision length is significantly shorter; In the HALS group, postoperative pain is less than with open surgery; In the HALS group, postoperative hospital stay is shorter than with open surgery
MeSH Terms: conditions — Pain, Postoperative; Splenomegaly

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
ABSTRACT

Background: Although there are some comparative studies between laparoscopy and hand-assisted laparoscopic splenectomy (HALS) in splenomegaly cases, there is no study of the differences between HALS and open splenectomy (OS). Our aim was to compare the HALS and OS techniques in splenomegaly cases.

Methods: This prospective study included 27 patients undergoing splenectomy for splenic disorders at the Department of General Surgery, Istanbul Medical Faculty between February 2007 and October 2007. OS was performed on 14 patients, and HALS was performed in the other 13 patients.

Key words: HALS, open splenectomy, splenomegaly

DETAILED DESCRIPTION:
The advent of laparoscopic surgery, increasing experience in its performance and advances in techniques and surgical devices have all greatly influenced general surgery. The usefulness of laparoscopic surgery has already been well proven in cholecystectomy, esophageal antireflux surgery, and splenectomy for benign diseases (1). Laparoscopy is also now gaining recognition for procedures accompanied by lymph node dissection, such as gastric and colorectal surgery (2, 3). The development of hand-assisted laparoscopic surgery (HALS) has also brought about improvements in regard to various disadvantages that have previously been associated with laparoscopic surgery, including lack of tactile sensation feedback, poor depth perception, lack of quick access in the event of unexpected hemorrhage, and difficulties with intracorporal suturing. Such improvements have enabled the performance of advanced laparoscopic surgery (4).

To solve the problems associated with a long learning curve and long operating times, hand ports have been introduced. Through the hand port, the surgeon's hand can be introduced into the abdomen while the pneumoperitoneum is preserved. The use of a hand port reduces operating time and shortens the learning curve (5). It has already been suggested that procedures requiring an incision to remove a specimen or organ are most suitable for HALS (6).

Laparoscopic splenectomy (LS) for the normal-sized spleen has been shown to be a safe procedure, resulting in short hospital stays, low postoperative pain scores, technical hurdles and, as a result, can be more difficult. LS has advantages over open splenectomy (7), and it is now considered by many surgeons to be the procedure of choice for normal-sized spleens. Splenectomy for giant spleens using solely laparoscopic approaches is feasible, but it can be time consuming and challenging to any surgeon despite his or her high level of experience with laparoscopy.

With increased splenic sizes, LS becomes more technically challenging, although the procedure is still feasible (8,5). Hand-assisted laparoscopic technique allows the surgeon to place one hand into the abdominal cavity while maintaining the pneumoperitoneum, recovering tactile sense and improving the accuracy of manipulation. This has been verified in various complicated laparoscopic procedures, including colectomies, nephrectomies, and hepatectomies. Based on these experiences, HALS may be well suited for the removal of splenomegaly when the final spleen weight is greater than 500 g (9).

It would be of interest to assess whether outcomes of the HALS hybrid technique approximate those obtained with laparoscopy or with the open approach. Since comparative studies between laparoscopy and HALS have been already carried out, we compared open splenectomy with HALS for splenomegaly cases. To our knowledge, this is the first prospective study to compare the results of HALS and OS.

MATERIALS AND METHODS

This prospective study included 27 patients undergoing splenectomy for splenic disorders at the Department of General Surgery, Istanbul Medical Faculty between February 2007 and October 2007. Patients were selected randomly according to numbers on a random table and assigned to one of the two different surgical procedures. Twenty-seven patients with splenomegaly and primary splenic tumors were included in the study. The patients were divided into two groups according to the surgical procedure performed: open splenectomy (Group 1 :OS, n=14) and hand-assisted laparoscopic splenectomy (Group 2:HALS, n=13). The study plan was reviewed and approved by our institutional ethical committee, and informed consent was obtained for all patients.

Non-Hodgkin lymphomas (n=11) were the main indication for splenectomy in this study. There were also rarely encountered primary splenic hemangiomas (n=2) (Table 1). Splenomegaly was identified clinically by palpation of the spleen below the coastal margin and/or by radiological examination of computerized tomography (CT) scans (15 cm or longer in craniocaudal diameter), with final intact splenic weight ≥ 500 g.

The study parameters included age, sex, the greatest splenic diameter, preoperative platelet count, preoperative hematocrit level and postoperative diagnosis. Body Mass Index (BMI) was calculated as the ratio of weight (kg) divided by height squared (m2). All the patients were evaluated with the American Society of Anesthesiology (ASA) score (10). Operative data included operative time as measured from first skin incision to the application of dressings, intraoperative blood loss, splenic weight after intact removal, conversion, pain score, and postoperative length of hospital stay. Complications were classified as intraoperative or postoperative. The pain of all patients was scored during postoperative days. The visual analogue scale defined by Wewers (11) was used for the evaluation of the degree of pain.

All the patients were vaccinated against pneumococci with Pneumovax 23 (Merck & Co Inc., Whitehouse Station, NJ, USA) two weeks before the operation. All patients received antibiotic prophylaxis (Sulbactam and ampicillin 1 g, intravenously). All patients received general anesthesia during surgery and a standardized analgesic regimen. HALS and OS were performed by the same surgical team. Post-operative analgesia was achieved by patient-controlled analgesia via a pump containing a standard narcotic analgesic solution. All patients received the same non-steroidal antinflammatory drug (lornoxicam 8 mg, twice a day, intravenously) and the same narcotic analgesic (pethidine 50 mg, twice a day, intramuscularly) on the first and second postoperative day.

Surgery Open Surgery(Group 1) Patients were placed in supine position. Since all patients had splenomegaly, preferred incisions were left subcostal. Only three patients requiring synchronous cholecystectomy had upper midline laparotomy incisions (18 cm, 18 cm and 20 cm in length). After routine whole abdominal exploration, with the assistance of abdominal retractors and the first assistance, the inferior pole and medial splenogastric ligament were dissected first, and then the splenorenal ligament and superior pole of the splenophrenic ligament were dissected. The LigaSure vessel sealing system (Valleylab division of Tyco Healthcare, Mansfield, MA) was used for the majority of the dissection. After this, the splenic vascular pedicule was separated from the pancreatic tail with careful dissection. In splenomegaly cases, if the splenic and perisplenic anatomy was appropriate, the ideal ligation of the splenic hilum was outside the abdomen (Figure 1). The splenic artery and splenic vein were ligated with silk (00) and sectioned. In the cases of massive splenomegaly, the main truncus of the splenic artery was ligated before the dissection to minimize blood loss and to allow the return of blood inside the spleen back to the circulation.

Figure 1- Splenic hilum ligation outside of the abdominal cavity

After the removal of the spleen, hemostasis was rechecked, and an aspirative drain was routinely placed. The abdominal wall was closed with loop polydioxanone (no: 1) in two layers with running sutures.

HALS procedure(Group 2) Patients were placed in a semilateral position with the left side elevated 30˚. The surgeon stood on the patients' right side with the camera operator. First, a hand port incision was made in the upper midline (Figure 2). The incision measured 7-8 cm (depending on the size of the surgeon's glove) in all cases. Then, the hand-assisted device Omniport (Advanced Surgical Concepts, Co. Wicklow, Ireland) was installed.

Figure 2- Omniport placed through an 8 cm upper midline incision in the HALS technique

The surgeon's left (non-dominant) hand was placed into the abdominal cavity through the device. The 10-mm 30˚ laparoscope was placed at the inferior or superior crease of the umbilicus depending on the spleen size and location. The 10-mm main operating port was in the midclavicular line at the level of the umbilicus. Carbon dioxide was insufflated continuously with 13 mmHg for constant pneumoperitoneum. An intraabdominal exploration for accessory spleen was the first step. LigaSure was used as above. With the assistance of the intraabdominal hand, the inferior pole and medial splenogastric ligament were dissected first, and then the splenorenal ligament and superior pole of the splenophrenic ligament were dissected. Then, the splenic vascular pedicule was separated from the pancreatic tail by finger dissection. The splenic artery and splenic vein were either ligated with LigaSure or silk (00) and sectioned or dissected with an endo vascular stapler (Endo-GIA).

In the cases of massive splenomegaly, the splenic artery was ligated before the dissection to gain enough operative space; this was also the case for LS. Finally, the spleen was placed into a retrieval bag and extracted intact via the hand port incision. Routinely, a suction drain was placed in the splenic fossa.

Statistical analysis Data are reported as the mean ± SD. The analysis was performed with the statistical package SPSS 10.1 (SPSS, Chicago, IL). Differences between variables were compared with nonparametric Mann Whitney-U and Student's t and chi-square tests. Spearman correlation analysis was performed for all patients. Results were considered statistically significant when the two-tailed p value was less than 0.05.

DISCUSSION

In 1991, Delaitre et al. attempted the first laparoscopic LS (12). Since then, the laparoscopic approach for splenectomy has gained wide acceptance and has been shown by several groups to be a technically successful, safe, and effective procedure. LS is now considered the standard approach to removing a normal-sized spleen for patients without other contraindications. In cases of splenomegaly, LS is also feasible in experienced hands, but, because the larger-sized spleen makes the operative space narrow, the exposure is limited, and manipulations are difficult, the LS procedure becomes more technically challenging. The hypervascularization and dense adhesions around the spleen hamper the surgeon's performance as well. Moreover, once the dissection is completed, the extraction of a giant spleen with a solely laparoscopic approach by placing it into a retrieval bag followed by morcellation can be difficult, and it can add considerable time to the procedure.

Some studies have suggested that LS for splenomegaly was associated with longer operation times, more blood loss, and higher intraoperative and postoperative complication rates than LS for normal-sized spleens (13). In addition, in some cases of splenomegaly, conversion is inevitable because of a requirement for an intact specimen for pathologic examination or because of serious hypervascularization and dense adhesion as the result of massive size (14, 15). Targarona et al. (14) indicated that the conversion rate was correlated with the spleen weight: for spleens weighing 400 - 1000 g, it was 0, but it rose to 25% for weights > 1000 g and to 75% for weights > 3000 g. In their LS group, conversions to laparoscopy-assisted splenectomy occurred in four patients (25%), including one case (spleen weight of 1600 g) for which pathologic examination determined a sarcoma and three cases of complicated procedures due to spleen weight > 3000 g (16). The median splenic weight in our HALS group was 800 (480-2110)g; we did not have any conversion to OS.

ELIGIBILITY:
Inclusion Criteria:

* Splenomegaly 15 cm or longer spleens
* Patient confirmation to join the study

Exclusion Criteria:

* Normal sized spleens
* Patient denial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with splenomegaly who will have splenectomy procedures either open or HALS
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UMUT BARBAROS, ASSIST.PROF, Principal Investigator — Istanbul Fcaulty of Medicine